CLINICAL TRIAL: NCT03371212
Title: A Prospective Randomized Trial of Modular Dual Mobility Acetabular Components Versus Conventional Single Bearing Components in Primary Total Hip Arthroplasty
Brief Title: A Prospective Randomized Controlled Trial of Dual-Mobility Components in Primary THA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17060804
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Serum Metal Levels, Specifically Cobalt, Chromium, and Titanium
Keywords: Dual Mobility; Serum metal levels

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 1 of 2 treatment groups, which they will be in for the duration of the study. Because of the nature of the study, there will be no crossover.
Who Masked: Participant
Masking Description: The patient will not have information about the treatment group they've been assigned to until after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Cohort (Active Comparator): Patients in this group will receive a Taperloc femoral stem, ceramic femoral head (size 32mm for acetabular components 48/50mm; size 36mm for acetabular components > 52mm), polyethylene bearing, and G7 acetabular shell.
  Interventions: Device: Conventional cohort
- Modular Dual Mobility Cohort (Experimental): Patients in this group will receive a Taperloc femoral stem, inner ceramic femoral head (28mm), mobile polyethylene bearing, cobalt alloy liner, and G7 acetabular shell.
  Interventions: Device: Dual mobility cohort

INTERVENTIONS:
Device: Dual mobility cohort — Patients will receive the Taperloc femoral stem, ceramic femoral head (size 32mm for acetabular components 48/50mm; size 36mm for acetabular components > 52mm), polyethylene bearing, and G7 acetabular shell.
  Arms: Modular Dual Mobility Cohort
Device: Conventional cohort — Patients will receive a Taperloc femoral stem, ceramic femoral head (size 32mm for acetabular components 48/50mm; size 36mm for acetabular components > 52mm), polyethylene bearing, and G7 acetabular shell
  Arms: Conventional Cohort

SUMMARY:
The aim of this study is to determine if the use of a modular dual mobility bearing is associated with clinically important increases in serum metal levels.

DETAILED DESCRIPTION:
Prosthetic dislocation following total hip arthroplasty (THA) remains a significant concern with a reported incidence of 0.2%-7.0% after primary and 10%-25% after revision THA. The risk of dislocation following THA is multifactorial and includes both surgeon-related factors (i.e. component positioning, surgical approach) and patient-related factors (i.e. gender, age). Dual mobility articulations have been shown to reduce the incidence of hip instability following THA. Dual mobility implants have been used in Europe for over 30 years, but have recently received an increased interest in the United States.

Initial dual mobility designs consisted of a cementless, monoblock acetabular component with a highly-polished metal inner bearing surface. Modular dual mobility prostheses have been introduced in which a modular cobalt-alloy liner is inserted into a hemispherical titanium acetabular component. Advantages of this construct include familiarity of use of a standard titanium acetabular component and the ability to use supplemental screw fixation. However, the potential for fretting corrosion between the cobalt-alloy liner and the titanium acetabular component remains a concern.

In a retrospective review of 100 consecutive patients undergoing primary THA using a modular dual mobility prosthesis, the authors found 21% of patients to have a serum cobalt level above the normal range, with 9% significantly above normal (> 1.6 ug/L), at a mean of 27.6 months postoperatively. In addition, a recent prospective cohort study of 26 patients receiving the same prosthesis showed elevated whole blood mean cobalt levels in patients receiving a modular dual mobility prosthesis versus patients receiving a conventional bearing (0.23 + 0.39 vs. 0.15 + 0.07ug/L, p<0.001) at 1 year postoperatively. Four patients in the dual mobility cohort had a whole blood cobalt level outside the reference range (maximum 1.81 ug/L).

To the investigators knowledge no prospective, randomized controlled trial has been performed comparing dual mobility bearings to a conventional single-bearing design. Therefore, the purpose of this study is to compare the use of a conventional single-bearing ceramic-on-polyethylene surface to use of a modular dual mobility bearing in a prospective, randomized controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Willingness to undergo serial postoperative venipuncture for serum meal analysis
* BMI < 40
* Patients that are eligible for the requisite implants as deemed by their surgeon

Exclusion Criteria:

* Clinically significant systemic chronic disease
* Diminished renal function
* Presence of any metal-containing implant outside of the oral cavity
* History of prior hip surgery involving an internal fixation device
* History of hip infection
* Preoperative diagnosis other than osteoarthritis
* Anticipated need for another joint replacement surgery within one year
* Patients taking chromium supplements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2035-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum chromium levels, measures chromium level in the serum in ug/L | up to 5 years
  Assays for each subject for serum chromium in ug/L
Serum cobalt levels, measures cobalt level in the serum in ug/L | up to 5 years
  Assays for each subject for serum cobalt in ug/L
Serum titanium levels, measures titanium level in the serum in ug/L | up to 5 years
  Assays for each subject for serum titanium in ug/L

SECONDARY OUTCOMES:
Patient reported outcome measures (survey) for SF-12 score. | up to 5 years
  Subjects will complete the industry common SF-12 survey and total score will be used. Higher scores are better, score of 100 is maximum.
Patient reported outcome measures (survey) for the Harris Hip Score | up to 5 years
  Subjects will complete the industry common Harris Hip survey and total score will be used. Higher scores are better, score of 100 is maximum.
Patient reported outcome measures (survey) for the Hoos Jr. score. | up to 5 years
  Subjects will complete the industry common HOOS Jr. survey and total score will be used. Higher scores are better, score of 100 is maximum.
Patient reported outcome measures (survey) for the SANE score. | up to 5 years
  Subjects will complete the the industry common SANE survey and total score will be used. Higher scores are better, score of 100 is maximum.
Patient reported outcome measures (survey) for the UCLA activity score. | up to 5 years
  Subjects will complete the the industry common UCLA survey and total score will be used. Higher scores are better, score of 100 is maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel PD, Potts A, Froimson MI. The dislocating hip arthroplasty: prevention and treatment. J Arthroplasty. 2007 Jun;22(4 Suppl 1):86-90. doi: 10.1016/j.arth.2006.12.111. PMID 17570285
- [Background] Berry DJ. Unstable total hip arthroplasty: detailed overview. Instr Course Lect. 2001;50:265-74. PMID 11372323
- [Background] Nam D, Salih R, Brown KM, Nunley RM, Barrack RL. Metal Ion Levels in Young, Active Patients Receiving a Modular, Dual Mobility Total Hip Arthroplasty. J Arthroplasty. 2017 May;32(5):1581-1585. doi: 10.1016/j.arth.2016.12.012. Epub 2016 Dec 21. PMID 28057394
- [Background] Haughom BD, Plummer DR, Moric M, Della Valle CJ. Is There a Benefit to Head Size Greater Than 36 mm in Total Hip Arthroplasty? J Arthroplasty. 2016 Jan;31(1):152-5. doi: 10.1016/j.arth.2015.08.011. Epub 2015 Aug 14. PMID 26360768
- [Background] Matsen Ko LJ, Pollag KE, Yoo JY, Sharkey PF. Serum Metal Ion Levels Following Total Hip Arthroplasty With Modular Dual Mobility Components. J Arthroplasty. 2016 Jan;31(1):186-9. doi: 10.1016/j.arth.2015.07.035. Epub 2015 Jul 23. PMID 26318084
- [Background] Heffernan C, Banerjee S, Nevelos J, Macintyre J, Issa K, Markel DC, Mont MA. Does dual-mobility cup geometry affect posterior horizontal dislocation distance? Clin Orthop Relat Res. 2014 May;472(5):1535-44. doi: 10.1007/s11999-014-3469-1. Epub 2014 Jan 24. PMID 24464508
- [Background] Langlais FL, Ropars M, Gaucher F, Musset T, Chaix O. Dual mobility cemented cups have low dislocation rates in THA revisions. Clin Orthop Relat Res. 2008 Feb;466(2):389-95. doi: 10.1007/s11999-007-0047-9. Epub 2008 Jan 10. PMID 18196422
- [Background] Loving L, Lee RK, Herrera L, Essner AP, Nevelos JE. Wear performance evaluation of a contemporary dual mobility hip bearing using multiple hip simulator testing conditions. J Arthroplasty. 2013 Jun;28(6):1041-6. doi: 10.1016/j.arth.2012.09.011. Epub 2013 Feb 22. PMID 23434106
- [Background] Civinini R, Carulli C, Matassi F, Nistri L, Innocenti M. A dual-mobility cup reduces risk of dislocation in isolated acetabular revisions. Clin Orthop Relat Res. 2012 Dec;470(12):3542-8. doi: 10.1007/s11999-012-2428-y. Epub 2012 Jun 15. PMID 22700131
- [Background] Hamadouche M, Arnould H, Bouxin B. Is a cementless dual mobility socket in primary THA a reasonable option? Clin Orthop Relat Res. 2012 Nov;470(11):3048-53. doi: 10.1007/s11999-012-2395-3. PMID 22639330
- [Background] Epinette JA, Beracassat R, Tracol P, Pagazani G, Vandenbussche E. Are modern dual mobility cups a valuable option in reducing instability after primary hip arthroplasty, even in younger patients? J Arthroplasty. 2014 Jun;29(6):1323-8. doi: 10.1016/j.arth.2013.12.011. Epub 2013 Dec 16. PMID 24444567
- [Background] Plummer DR, Christy JM, Sporer SM, Paprosky WG, Della Valle CJ. Dual-Mobility Articulations for Patients at High Risk for Dislocation. J Arthroplasty. 2016 Sep;31(9 Suppl):131-5. doi: 10.1016/j.arth.2016.03.021. Epub 2016 Mar 17. PMID 27101771
- [Background] McArthur BA, Nam D, Cross MB, Westrich GH, Sculco TP. Dual-mobility acetabular components in total hip arthroplasty. Am J Orthop (Belle Mead NJ). 2013 Oct;42(10):473-8. PMID 24278908
- [Background] Farizon F, de Lavison R, Azoulai JJ, Bousquet G. Results with a cementless alumina-coated cup with dual mobility. A twelve-year follow-up study. Int Orthop. 1998;22(4):219-24. doi: 10.1007/s002640050246. PMID 9795807